CLINICAL TRIAL: NCT03168477
Title: Electric Dry Needling and Spinal Manipulation vs. Impairment-based Mobilization, Exercise and Interferential Electrotherapy for Patients With Shoulder Impingement (Subacromial Pain Syndrome): a Multi-center Randomized Control Trial
Brief Title: Dry Needling and Manipulation vs. Mobilization, Exercise and Interferential Electrotherapy for Shoulder Impingement (Subacromial Pain Syndrome)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, Primary Investigator and President of Spinal Manipulation Institute and Dry Needling Institute of the American Academy of Manipulative Therapy, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT0012
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Subacromial Pain Syndrome
MeSH Terms: interventions — Dry Needling; Manipulation, Spinal; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry needling and spinal manipulation (Experimental)
  Interventions: Other: dry needling; Other: spinal manipulation
- mobilization, exercise, modalities (Active Comparator)
  Interventions: Other: mobilization; Other: exercise; Other: modalities

INTERVENTIONS:
Other: dry needling — Dry needling to the supraspinatus (proximal/distal teno-osseus junction and musculotendinous junction under acromion process), deltoid muscle, upper trapezius muscle and levator scapulae muscle on the painful side. Clinicians may also needle the terres major, infraspinatous, rhomboids and thoracic paraspinals, as needed. Up to 12 treatment sessions over 6 weeks.
  Arms: dry needling and spinal manipulation
Other: spinal manipulation — HVLA thrust manipulation to cervical, thoracic and/or upper rib articulation (R1-R3).
  Arms: dry needling and spinal manipulation
Other: mobilization — Impairment-based mobilization targeting the muscles, scapulae and joint capsule of the painful shoulder. Up to 12 treatment sessions over 6 weeks.
  Arms: mobilization, exercise, modalities
Other: exercise — Impairment-based exercise targeting the muscles, scapulae and joint capsule of the painful shoulder. Up to 12 treatment sessions over 6 weeks.
  Arms: mobilization, exercise, modalities
Other: modalities — Interferential electrotherapy targeting the muscles, scapulae and joint capsule of the painful shoulder. Up to 12 treatment sessions over 6 weeks.
  Arms: mobilization, exercise, modalities

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with shoulder impingement (subacromial pain syndrome): electric dry needling and spinal manipulation versus impairment-based mobilization, exercise, and interferential electrotherapy. Physical therapists commonly use all of these techniques to treat shoulder impingement (subacromial pain syndrome). This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patients with shoulder impingement (subacromial pain syndrome) will be randomized to receive 2 treatment sessions per week for up to 6 weeks (up to 12 sessions total) of either: (1) electric dry needling and spinal manipulation or (2) impairment-based mobilization, exercise and interferential electrotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult over the age of 18 years old that is able to read, write and speak English
2. Primary complaint of anterolateral shoulder pain lasting longer than 6 weeks
3. One or more of the following special tests:

   1. Positive Neer Impingement test-i.e. pain with passive overpressure at full shoulder flexion with the scapula stabilized.
   2. Positive Hawkins-Kennedy test-i.e. pain with passive internal rotation at 90° of shoulder and elbow flexion
4. Pain with ONE or more of the following active movements and resisted isometric tests

   1. Pain with active shoulder elevation
   2. Pain with resisted shoulder external rotation at 90 deg of abduction
   3. Pain with resisted shoulder abduction in Empty Can Test positon - i.e. 90 deg of shoulder abduction, 30 deg of horizontal adduction (i.e. in scapular plane) and full internal rotation (i.e. thumb down)

Exclusion Criteria:

1. Report of red flags to manual physical therapy to include: severe hypertension, infection, uncontrolled diabetes, peripheral neuropathy, heart disease, stroke, chronic ischemia, edema, severe varicosities, tumor, metabolic disease, prolonged steroid use, fracture, RA, osteoporosis, severe vascular disease, malignancy, etc.
2. History of shoulder injection within the past 3 months.
3. History of shoulder dislocation, subluxation, fracture, adhesive capsulitis, or cervical, thoracic or shoulder surgery.
4. Isolated acromioclavicular joint pathology (i.e. the only location of symptoms is localized specifically with one finger directly over the acromioclavicular joint and nowhere else, and reproduced only with acromioclavicular palpation by the examiner.)
5. Evidence of cervical radiculopathy, radiculitis or referred pain from the c-spine
6. Full-thickness rotator cuff tears (evidenced by MRI and/or positive lag signs)
7. Baseline SPADI of not less than 20%
8. History of breast cancer on involved side.
9. Prior treatments (eg. Acupuncture, physical therapy, chiropractic, dry needling, massage therapy, injections) to the involved limb over past 3 months.
10. Pending litigation for an injury.
11. Psychiatric disorders or cognitively impaired
12. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Pain (NPRS) (Rating Score) | baseline, 2-weeks, 4-weeks, 3 months
  Rating Score. Baseline score must exceed 2/10 to be included in the study.
Change in Shoulder Pain and Disability Index | baseline, 2-weeks, 4-weeks, 3 months
  The SPADI Pain subscale is measured on a 0-130 scale. Greater scores indicate increased pain. Patient must have score of 20% or greater to participate in study on both the pain and disability section.

SECONDARY OUTCOMES:
Change in Global Rating of Change Score | 2 week, 4 weeks, 3 months
Change in Medication Intake (Frequency of medication intake in last week) | baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Evolution Sports Physiotherapy, Cockeysville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided